CLINICAL TRIAL: NCT03840733
Title: Linking Temporal Patterns of Modifiable Behaviors to Weight Loss Outcomes
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 18-1319; K01HL145023 (NIH)
Record Dates: First submitted 2019-01-29; First posted 2019-02-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Weight Change, Body
Keywords: physical activity; sleep; eating patterns; energy expenditure
MeSH Terms: conditions — Obesity; Body Weight Changes; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants from NCT01985568 or NCT03411356: All subjects who previously enrolled in the Parent Study's behavioral weight loss intervention (NCT01985568 or NCT03411356).

SUMMARY:
This study is designed as an observational trial. The objective of this study is to follow-up with participants 3 years after completion of an 18-month comprehensive behavioral weight loss intervention. Outcomes of interest include change in body weight, body composition, physical activity, energy intake, and sleep. In addition, investigators will explore the associations between current physical activity, sleep, and energy intake patterns and body weight regulation.

DETAILED DESCRIPTION:
A total of 170 participants were initially enrolled in the comprehensive behavioral weight loss intervention.In this study, investigators will conduct a follow-up visit 3 years after the completion of the intervention. Only participants who completed the behavioral weight loss intervention will be enrolled in this study. Participants will undergo testing of body weight, body composition, physical activity patterns, energy intake patterns, sleep patterns, resting metabolic rate, and total daily energy expenditure.

ELIGIBILITY:
Inclusion Criteria:

* Previous enrollment in standard behavioral weight loss intervention (NCT01985568 or NCT03411356)
* Age 20-60 (This age range has been selected based upon the participants enrolled in the Parent Trial)
* Capable and willing to give informed consent
* Possess a smartphone to install and utilize the meal timing application
* Capable and willing to wear the Actigraph, ActivPAL and Actiwatch-2 for 24 hours/day for 28 consecutive days
* Willing to complete the Total Daily Energy Expenditure (TDEE) assessment which includes multiple urine collections and drinking stable water isotopes

Exclusion Criteria:

* Being considered unsafe to participate as determined by the study physician (Dr. Catennaci)
* New diagnosis of a medical condition (not observed in the Parent Trial) which may affect weight or energy metabolism (e.g. depression, CVD, diabetes, uncontrolled hypertension, untreated thyroid, renal, hepatic diseases)
* Women who became pregnant after completing the Parent Trial
* Current use or use within the last 6 months of prescription or over-the-counter medications known to affect appetite, weight, and sleep

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants previously enrolled in an 18-month behavioral weight loss intervention at the University of Colorado Anschutz Medical Campus. (NCT01985568)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Weight Change | Baseline to 54 months
  Change in body weight (kg)
Weight Maintenance | 18 months to 54 months
  Change in body weight (kg)
Fat Mass Change | Baseline to 54 months
  Change in Fat Mass (kg)
Fat Free Mass Change | Baseline to 54 months
  Change in Fat Free Mass (kg)
Fat Mass Maintenance | 18 months to 54 months
  Change in Fat Mass (kg)
Fat Free Mass Maintenance | 18 months to 54 months
  Change in Fat Free Mass (kg)

SECONDARY OUTCOMES:
Change in Physical Activity Patterns | 0, 6, 12, 18, 24, 54 month
  Physical activity patterns as measured by SenseWear armband (min/day)
Physical Activity Patterns | 54 month
  Physical activity patterns as measured by ActivPAL, Actigraph (min/day)
Change in Sleep | 0, 6, 12, 18, 24, 54 month
  Sleep patterns as measured by SenseWear armband (h/day)
Sleep Patterns | 54 month
  Sleep patterns as measured by Actiwatch-2, ActivPAL, Actigraph (h/day)
Change in Energy Intake | 0, 6, 12, 18, 54 month
  Energy Intake patterns as measured by 3 day food record (kcal/day
Energy Intake Patterns | 54 month
  Energy Intake patterns as measured by 24 hour food recall and meallogger smartphone application (kcal/day)
Resting Metabolic Rate | 54 month
  Resting metabolic rate as measured using indirect calorimetry (kcal/day)
Total Daily Energy Expenditure | 54 month
  Total Daily Energy Expenditure as measured by doubly labeled water (kcal/day)
Physical Activity Energy Expenditure | 54 month
  Physical Activity Energy Expenditure as measured by doubly labeled water (kcal/day)

CONTACTS AND LOCATIONS:
Overall Officials: Seth A Creasy, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No